CLINICAL TRIAL: NCT02754362
Title: A Toll-like Receptor Agonist as an Adjuvant to Tumor Associated Antigens (TAA) Mixed With Montanide ISA-51 VG With Bevacizumab for Patients With Recurrent Glioblastoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to personnel changes / departure of Dr. Chi.
Sponsor: NYU Langone Health (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15-00044
Record Dates: First submitted 2016-04-13; First posted 2016-04-28 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Glioblastoma; Glioma
Keywords: Poly-ICLC and bevacizumab; humanized monoclonal antibody
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Bevacizumab; poly ICLC; Protein Subunit Vaccines; Adjuvants, Immunologic; keyhole-limpet hemocyanin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Block 1 (Experimental)
  Interventions: Drug: Bevacizumab
- Block 2 (Experimental)
  Interventions: Drug: Bevacizumab; Biological: Peptide Vaccine; Drug: Poly-ICLC as immune adjuvant; Drug: Keyhole limpet hemocyanin (KLH)
- Block 3 (Experimental)
  Interventions: Drug: Bevacizumab; Biological: Peptide Vaccine; Drug: Poly-ICLC as immune adjuvant

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab is a humanized monoclonal antibody that targets vascular endothelial growth factor (VEGF), a proangiogenic factor which aids in tumor vessel formation.
  Other Names: Hiltonol®
Biological: Peptide Vaccine — Vaccine of long synthetic peptides encoding T cell epitopes in tumor associated antigens.
  Vaccine Consists of:
  EGFRvIII peptide 100 mcg IL13Ralpha peptide 100 mcg EphA2 peptide 100 mcg Her2/neu peptide 100 mcg YKL-40 peptide 100 mcg
  Arms: Block 2; Block 3
Drug: Poly-ICLC as immune adjuvant — Poly-ICLC is a toll like receptor 3 agonist which directly activates dendritic cells and triggers natural killer cells to kill tumor cells.
  Arms: Block 2; Block 3
Drug: Keyhole limpet hemocyanin (KLH) — Potent Immunogen used in vaccine approaches for a number of diseases including cancer, AIDS, and infectious diseases
  Arms: Block 2

SUMMARY:
This is a phase II study to determine the immunogenicity and efficacy of a vaccine composed of tumor associated long synthetic peptides mixed with Montanide ISA-51 VG administered with polyinosinic-polycytidylic acid - poly-L-lysine carboxymethylcellulose (Poly-ICLC) and bevacizumab in adults with recurrent glioblastoma.

DETAILED DESCRIPTION:
All patients will receive the same dose of vaccine, Poly-ICLC and bevacizumab. The therapy consists of 3 blocks. During the first block, patients will receive bevacizumab every 2 weeks for 2 doses. During block 2, patients will receive vaccine + Poly-ICLC + bevacizumab on weeks 1, 3, 5 and 7. An MRI will be performed after week 7 therapy. If there is no significant progression, then the patients will continue with block 3. During block 3, therapy consists of vaccine + Poly-ICLC monthly and bevacizumab every 2 weeks for 10 months. Keyhole limpet hemocyanin (KLH) will be given as a positive control with the first vaccine. Immune studies will be performed in all patients enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Disease Status. Patients with first recurrence of glioblastoma (WHO IV). Patients must have histological confirmation of glioblastoma (WHO grade IV) either at diagnosis or at first recurrence. Patients with diffuse intrinsic pontine glioma (DIPG) are not eligible.
* Karnofsky performance status > 50. Patients who are unable to walk because of paralysis but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Adequate organ function:

Hematologic: absolute lymphocyte count > 200/mm3 Platelets > 100,000 Hepatic:AST/ALT < 5 x the upper limit of institutional normal Total bilirubin < 1.5 x the upper limit of institutional normal Renal: serum creatinine < 1.5 mg/ml; Urine protein/creatinine ratio < 2.0 at screening Cardiac: Hypertension must be well controlled on stable doses of medication. BP must be < 140/90.

* Life expectancy >3 months
* Patients must have fully recovered from previous surgery, chemotherapy, radiotherapy and biologic therapy. No surgery, chemotherapy, radiation therapy or immunotherapy within 4 weeks prior to the first dose of study agent or bevacizumab (6 weeks for nitrosureas).
* Patients must have no measurable disease or minimal residual disease defined as <1.5cm2 enhancement. Patients may have surgery to achieve < 1.5cm2 residual.
* Tumor tissue must be available either from initial diagnosis or relapse for testing of antigen expression.
* Informed consent must be signed by the patient. Individuals who lack capacity to sign consent will be excluded. Patients must be able to read and/or understand the details of the study and provide written evidence of informed consent as approved by the IRB.

Exclusion Criteria:

* Serious illness, such as uncontrolled infections requiring antibiotics
* History of immunodeficiency disease (such as HIV) or autoimmune disease except vitiligo
* Concomitant treatment with systemic dexamethasone (or it's equivalent) greater than 2mg/day. Topical (but not at the proposed vaccination site) or inhalational steroids are permitted
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior the first dose of study agent.
* Pregnant or lactating women are not permitted.
* Women of child-bearing potential not using medically acceptable means of contraception.
* Prior vaccine therapy for high grade glioma is not allowed.
* Other malignancy within 3 years prior to entry into the study, except for treated early-stage melanoma or non-melanoma skin cancer, or cervical carcinoma in situ
* Significant bleeding history
* Patients with serious or non-healing wound, ulcer, or bone fractures are not eligible.
* Patients must not have a history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to study entry.
* Patients must not have a known bleeding diathesis or coagulopathy.
* Patients must not have had significant vascular disease (eg, aortic aneurysm requiring surgical repair, deep venous or arterial thrombosis) within the last 6 months prior to study entry.
* Patients must not have evidence of new CNS hemorrhage on baseline MRI obtained within 14 days prior to study enrollment.
* Patients must not have a known thrombophilic condition (i.e. protein S, protein C or antithrombin III deficiency, Factor V Leiden, Factor II G20210A mutation, homocysteinemia or antiphospholipid antibody syndrome). Testing is not required in patients without thrombophilic history.
* Patients must not have a history of stroke, myocardial infarction, transient ischemic attack (TIA), severe or unstable angina, peripheral vascular disease, or grade II or greater congestive heart failure within the past 6 months prior to study entry.
* Patients must not have serious and inadequately controlled cardiac arrhythmias.
* Patients must not have a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the first dose of bevacizumab or anticipation of need for major surgical procedure during the course of the study.
* Patients must not have minor surgical procedures, fine needle aspirations, or core biopsies within 7 days prior to study enrollment.
* Patients with organ allografts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Assays to determine immunity to the vaccine's antigen | 9 Weeks
Measure of Humoral Immune Responses measured by ELISA | 9 Weeks
Antigen specific CD4+ and CD8+ T-cell reactivity to the peptide antigens measured by intracellular cytokine staining | 9 Weeks
  Measured either ex-vivo (assayed directly from thawed PBMCs) or following in-vitro pre-sensitization.
CD4+ and CD8+ T cell reactivity to KLH measured by T cell proliferation quantified by tritiated thymidine incorporation | 9 Weeks
Measure of Tumor Responses measured by the Response Evaluation Criteria in Solid Tumors (RECIST). | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Gardner, MD, Principal Investigator — New York University Medical School
Locations (1):
- NYU Perlmutter Cancer Center, New York, New York, United States